CLINICAL TRIAL: NCT07020403
Title: Development and Evaluation of a Mindfulness-Based on Emotional Eating Reduction Program
Brief Title: Mindfulness-Based Emotional Eating Intervention Program
Acronym: MB-EER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: tuğba çolak (Other)
Responsible Party: Sponsor-Investigator, tuğba çolak, ASSOC. PROFESSOR, Duzce University
Organization: Duzce University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DU-MBEER-2024
Record Dates: First submitted 2025-05-09; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Emotional Eating
Keywords: Emotional Eating; Mindfulness; Emotional Appetite; Mindful Eating
MeSH Terms: conditions — Emotional Eating

STUDY DESIGN:
Intervention Model Description: This study was conducted using a parallel-group experimental design with random assignment. Participants were divided into an intervention group and a control group. The intervention group received a 7-week Mindfulness-Based Emotional Eating Reduction (MB-EER) Program, while the control group received no intervention. Assessments were conducted at pre-test, post-test, and 3-month follow-up.
Who Masked: Participant
Masking Description: Only participants were blinded to their group assignment. The investigator and outcomes assessor were aware of group allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MB-EER Intervention Group (Experimental): Participants in this group received the 7-week Mindfulness-Based Emotional Eating Reduction (MB-EER) Program. The intervention was delivered online via Zoom and included weekly 2-hour sessions focusing on mindful eating practices, emotional regulation, and body awareness.
  Interventions: Behavioral: Mindfulness-Based Emotional Eating Reduction Program (MB-EER)
- Assessment-Only Control Group (No Intervention): Participants in this group received no intervention during the study period. They completed the same assessments at baseline, post-test, and 3-month follow-up as the intervention group.

INTERVENTIONS:
Behavioral: Mindfulness-Based Emotional Eating Reduction Program (MB-EER) — The MB-EER program was delivered to participants in the intervention arm over 7 weeks. Each session lasted 2 hours and was conducted weekly via Zoom. Participants attended in small groups, and sessions were led by trained facilitators. The intervention focused on guided mindfulness practices, mindful eating exercises, and group discussions.
  Other Names: MB-EER
  Arms: MB-EER Intervention Group

SUMMARY:
This study aims to develop and evaluate the effectiveness of a mindfulness-based intervention program called the Mindfulness-Based Emotional Eating Reduction (MB-EER) Program. The program is designed to reduce emotional eating behaviors in adults. Participants were randomly assigned to either an intervention group or a control group. The intervention group attended a 7-week online program with weekly sessions that included psychoeducation, mindfulness exercises (such as body scan and breath awareness), experiential activities, and group discussions. Data were collected at three time points: before the intervention, after the 7th week, and at a 3-month follow-up. Emotional eating, mindful eating, and emotional appetite levels were measured. Results showed that the MB-EER program effectively reduced emotional eating and emotional appetite while increasing mindful eating.

DETAILED DESCRIPTION:
This study aims to develop and evaluate a mindfulness-based intervention program (MB-EER) designed to reduce emotional eating behavior. The program was structured based on needs analyses conducted with experts and individuals with emotional eating experiences.

The MB-EER Program consists of 7 weekly sessions, each lasting approximately 2 hours, conducted online. Each session includes psychoeducational content, mindfulness-based practices (e.g., breath awareness, body scan), experiential activities, and group sharing.

Session Overview:

Focus on How You Eat - Differentiating emotional eating from physical hunger; raisin exercise

Recognizing Autopilot - Emotional triggers and automatic eating behaviors

Attention to Cues - Internal and external stimuli influencing eating behavior

Hunger and Fullness Signals - Awareness of body signals; water-drinking practice

Body Awareness and Self-Compassion - Developing supportive attitudes toward the body

Cultural Beliefs and Eating History - Social rules and learned eating habits

Maintenance and Reflection - Ensuring sustainability of skills, personal awareness

Research Design:

This study used a mixed-methods design, including both the development and experimental evaluation of the program:

Program Development Phase

Experimental Evaluation Phase

Quantitative design:

The experimental phase used a true experimental pre-test-post-test-follow-up control group design. Qualitative data were embedded throughout the process using semi-structured forms.

Participant Selection and Assignment:

Out of 135 initial applicants, Emotional Eating Scale (EES) scores were calculated and converted into Z scores using SPSS, since the scale lacks a clinical cut-off. 91 participants falling within ±2 SD were considered eligible and assessed for exclusion criteria.

8 individuals were excluded due to diagnosed eating disorders (e.g., bulimia, binge eating)

12 were excluded due to chronic conditions affecting appetite regulation (e.g., Hashimoto's, diabetes, thyroid)

2 individuals could not commit to the program

From the remaining 69 eligible participants, 40 were randomly assigned into experimental and control groups (20 each). However, due to dropouts during the process:

15 participants in the experimental group

15 participants in the control group completed the full study process and provided data at all time points.

Implementation:

The MB-EER program was delivered to the experimental group by the lead researcher.

Sessions were held online (Zoom) over 7 weeks, once per week.

The control group received no intervention.

All participants completed measurements at three points:

Pre-test (before the intervention)

Post-test (end of Week 7)

Follow-up test (3 months later)

Data Collection Instruments:

Emotional Eating Scale (EES-30)

Mindful Eating Scale (MES-30)

Emotional Appetite Questionnaire (EAQ-22)

Data Analysis:

Quantitative data were analyzed using SPSS v26.0

Parametric tests were used as normality assumptions were met

Statistical procedures included:

Two-factor mixed ANOVA

Wilks' Lambda multivariate repeated measures (MANOVA)

Bonferroni-adjusted pairwise comparisons

Qualitative data were evaluated using content and descriptive analysis

Findings:

The main hypothesis of the study was that the MB-EER Program is effective in reducing emotional eating and emotional appetite and improving mindful eating. This hypothesis was tested by comparing pre-, post-, and follow-up scores between experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older

Individuals reporting high levels of emotional eating

Willingness to participate in a 7-week online intervention program

Access to a computer and stable internet connection

Completion of informed consent form

Exclusion Criteria:

* Current diagnosis of an eating disorder (e.g., bulimia nervosa, binge eating disorder)

Diagnosis of a chronic medical condition that affects appetite (e.g., diabetes, thyroid disorders such as Hashimoto's disease)

Pregnancy

Inability to commit to regular attendance in the 7-week program

Participation in another psychological intervention during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Change in Emotional Eating Score (EES-30) from Baseline to Follow-up | Change from Baseline (Week 0) to Post-test (Week 7) and Follow-up (Week 12)
  The scale developed by Bilgen (2018) was adapted to reveal the relationship between emotions and eating. The scale consists of 4 sub-dimensions (Eating in Tense Situations, Eating to Cope with Negative Emotions, Self-Control, and Control in the Face of Stimuli). The scale is scored on a 5-point Likert scale, and the items consist of "Never (1)", "Rarely (2)", Sometimes (3)", 'Often (4)' and 'Always (5)' options. Both the sub-dimensions and the whole scale give a total score, and it is concluded that the higher the score obtained from the scale, the higher the emotional eating tendencies. The highest score that can be obtained from the scale is 150, and the lowest score is 30. The scale has a total of 30 items and three reverse-coded items. The Cronbach's Alpha internal consistency coefficient of the scale for this study was calculated as .92.
Mindful eating questionnaire (MEQ-30) | Change from Baseline (Week 0) to Post-test (Week 7) and Follow-up (Week 12)
  The Mindful Eating Questionnaire (MEQ) is a 30-item self-report scale adapted to Turkish by Köse et al. (2016). It includes seven subscales: Disinhibition, Emotional Eating, Eating Control, Focusing, Eating Discipline, Mindfulness, and Interference. Items are rated on a 5-point Likert scale (1 = Never, 5 = Always). Higher scores indicate greater mindful eating. Twenty items are reverse-coded. Cronbach's alpha = .72.
Emotional appetite questionnaire (EAQ-22) | Change from Baseline (Week 0) to Post-test (Week 7) and Follow-up (Week 12)
  The Emotional Appetite Questionnaire (EAQ-22), validated in Turkish by Demirel et al. (2014), is a 22-item self-report scale assessing appetite changes in response to emotional states and situations. Items are rated from 1 to 9: 1-4 = less appetite, 5 = no change, 6-9 = more appetite. Subscales include emotions (14 items) and situations (8 items), each split into positive and negative categories. Higher scores indicate greater emotional appetite. Cronbach's alpha = .71.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Seda Çolak Turan, Principal Investigator — tugbacolak@duzce.edu.tr
Locations (1):
- Duzce University, Düzce, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) will be shared, including raw scores from the Emotional Eating Scale (EES-30), Mindful Eating Scale (MES-30), and Emotional Appetite Questionnaire (EAQ-22) collected at three time points (pre-test, post-test, and 3-month follow-up). Data will be available to qualified researchers upon request via Open Science Framework at [https://osf.io/u3wqk/].
Supporting Information: SAP, CSR
Time Frame: Individual participant data (IPD) has been available since December 8, 2024, and will remain available until December 8, 2029.
Access Criteria: Qualified researchers who provide a methodologically sound proposal will be granted access to the deidentified individual participant data (IPD). Data includes scores from the Emotional Eating Scale (EES-30), Mindful Eating Scale (MES-30), and Emotional Appetite Questionnaire (EAQ-22) at baseline, post-test, and follow-up. Requests should be submitted via the Open Science Framework (https://osf.io/yk3mp/) platform. Access will be granted for research purposes only and in compliance with data use agreements.
URL: https://osf.io/u3wqk/

REFERENCES:
- See also: Project page for the "Mindfulness-Based Emotional Eating Reduction (MB-EER) Program" including study protocol, data sharing plan, and materials. — https://osf.io/u3wqk/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT07020403/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT07020403/ICF_001.pdf